CLINICAL TRIAL: NCT04301076
Title: A Phase 1 Study of Lenalidomide in Combination With EPOCH Chemotherapy for HTLV-Associated Adult T-Cell Leukemia-Lymphoma (ATLL)
Brief Title: Testing the Addition of an Anti-cancer Drug, Lenalidomide, to the Usual Combination Chemotherapy Treatment ("EPOCH") for Adult T-Cell Leukemia-Lymphoma (ATLL)
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Other - Pending amendment.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-01535; NCI-2020-01535 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10335 (Other: Yale University Cancer Center LAO); 10335 (Other: CTEP); UM1CA186689 (NIH); UM1CA186704 (NIH)
Record Dates: First submitted 2020-03-06; First posted 2020-03-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Adult T-Cell Leukemia/Lymphoma; Adult T-Cell Leukemia/Lymphoma; Chronic Adult T-Cell Leukemia/Lymphoma; HTLV-1 Infection
MeSH Terms: conditions — Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; HTLV-I Infections | interventions — Specimen Handling; Biopsy; Cyclophosphamide; Doxorubicin; Etoposide; Lenalidomide; Magnetic Resonance Spectroscopy; Prednisone; deltacortene; prednylidene; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (lenalidomide, EPOCH) (Experimental): INDUCTION THERAPY: Patients receive lenalidomide PO QD on days 1-14 of 21 day cycles or days 1-21 or 1-28 of 28 day cycles. Patients receive doxorubicin hydrochloride IV continuously on days 1-4, vincristine sulfate IV continuously on days 1-4, etoposide IV continuously on days 1-4, prednisone PO on days 1-5, and cyclophosphamide IV over 1-4 hours on day 5. Treatment repeats every 21 or 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients with CR, PR, or SD may receive up to 2 additional cycles of lenalidomide, doxorubicin hydrochloride, vincristine sulfate, etoposide, prednisone, and cyclophosphamide at the discretion of the investigator and/or up to an additional 2 years of lenalidomide in the absence of disease progression or unacceptable toxicity.
  Patients undergo bone marrow biopsy at baseline and as clinically indicated. Patients undergo PET/CT or CT, tissue and blood sample collection throughout.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Lenalidomide; Procedure: Positron Emission Tomography; Drug: Prednisone; Drug: Vincristine Sulfate

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo tissue and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo PET/CT or CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase I trial studies the side effects and best dose of lenalidomide when given together with usual combination chemotherapy (etoposide, prednisone, vincristine sulfate [Oncovin], cyclophosphamide, and doxorubicin hydrochloride [hydroxydaunorubicin hydrochloride], or "EPOCH") in treating adult T-cell leukemia-lymphoma. Lenalidomide may help shrink or slow the growth of adult T-cell leukemia-lymphoma. Drugs used in chemotherapy, such as etoposide, vincristine, cyclophosphamide, and doxorubicin, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Anti-inflammatory drugs such as prednisone lower the body's immune response and are used with other drugs in the treatment of some types of cancer. Giving lenalidomide and the usual combination chemotherapy may work better in treating adult T-cell leukemia-lymphoma compared to the usual combination chemotherapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safest and most tolerable dose and schedule of lenalidomide to combine with etoposide, prednisone, vincristine sulfate (Oncovin), cyclophosphamide, and doxorubicin hydrochloride (hydroxydaunorubicin hydrochloride) (EPOCH) chemotherapy in adult T-cell leukemia-lymphoma (ATL/ATLL).

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To determine if lenalidomide and EPOCH activity results in significant improvement in remission rates, duration of remissions, and overall survival (OS) as compared to historical controls.

III. To determine if lenalidomide and EPOCH activity correlates with T-cell receptor (TCR) pathway gene mutational spectrum.

IV. To determine effects of lenalidomide and EPOCH on human T-cell leukemia virus type 1 (HTLV-1) proviral deoxyribonucleic acid (DNA) and ribonucleic acid (RNA) loads.

V. To determine effects of lenalidomide and EPOCH on HTLV-1 clonality.

OUTLINE: This is a dose-escalation study of lenalidomide followed by a dose-expansion study.

INDUCTION THERAPY: Patients receive lenalidomide orally (PO) once daily (QD) on days 1-14 of 21 day cycles or days 1-21 or 1-28 of 28 day cycles. Patients receive doxorubicin hydrochloride intravenously (IV) continuously on days 1-4, vincristine sulfate IV continuously on days 1-4, etoposide IV continuously on days 1-4, prednisone PO on days 1-5, and cyclophosphamide IV over 1-4 hours on day 5. Treatment repeats every 21 or 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients with complete response (CR), partial response (PR), or stable disease (SD) may receive up to 2 additional cycles of lenalidomide, doxorubicin hydrochloride, vincristine sulfate, etoposide, prednisone, and cyclophosphamide at the discretion of the investigator and/or up to an additional 2 years of lenalidomide in the absence of disease progression or unacceptable toxicity.

Patients undergo bone marrow biopsy at baseline and as clinically indicated. Patients undergo positron emission tomography/computed tomography (PET/CT) or CT, tissue and blood sample collection throughout the trial.

After completion of study treatment, patients are followed up for 2 years from end of induction. Patients who do not continue on lenalidomide maintenance are followed every 3 months for up to 2 years from the end of induction, progression, withdrawal, or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed CD2+, CD3+, or CD4+ acute, lymphoma or poor-risk chronic subtypes of ATLL including previously untreated or previously treated individuals who have received no more than 1 previous cycle of EPOCH, cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP), or cyclophosphamide, doxorubicin, vincristine, prednisone, and etoposide (CHOPE)
* Patients previously treated with azidothymidine (AZT), interferon (IFN), bexarotene, or mogamulizumab are eligible. Patients with stable disease at high risk of relapse from prior non-combination chemotherapy containing treatment are eligible to participate
* Documentation of HTLV infection by enzyme-linked immunosorbent assay (ELISA) in individuals with confirmation of HTLV-1 infection (by immunoblot or polymerase chain reaction [PCR]) or a consistent clinical picture (including two of three of: 1) CD4+ leukemia or lymphoma, 2) hypercalcemia, and/or 3) Japanese, Caribbean, or South American birthplace) is required for enrollment. Confirmation of HTLV-1 infection is required to continue the subject on protocol after the first cycle of therapy. Patients will be enrolled based on reports from local or referral labs (e.g., Mayo Clinic or LabCorp). Confirmation will be performed by Ratner Lab at Washington University, retrospectively, but this is not a Clinical Laboratory Improvement Amendments (CLIA) assay and is not reimbursed by insurance
* Age ≥ 18 years

  * Because no dosing or adverse event (AE) data are currently available on the use of lenalidomide in combination with EPOCH in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,000/mm^3 unless decreased due to bone marrow (BM) involvement with lymphoma
* Platelets >= 100,000/mm^3 unless decreased due to BM involvement with lymphoma
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN), if potentially due to lymphoma, in the dose-expansion cohort, the first cycle may be given without lenalidomide and if transaminitis and bilirubinemia improves to meet parameters, participant may be enrolled
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2 x institutional ULN, if potentially due to lymphoma, in the dose-expansion cohort, the first cycle may be given without lenalidomide and if transaminitis and bilirubinemia improve to meet parameters, participant may be enrolled
* Creatinine =< institutional ULN OR glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patients must have a life expectancy > 12 weeks
* Patients must have no serious active infection requiring therapy at the time of study entry
* Patients must not require the concurrent use of chemotherapy, interferon, zidovudine, arsenic, radiation therapy, or other specific anti-tumor therapy, during the course of this study
* The effects of lenalidomide on the developing human fetus are unknown. Immunodulatory derivative (immunomodulatory imide drug [IMiD]) agents as well as other therapeutic agents used in this trial are known to be teratogenic. Females of child-bearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days prior to, and again within 24 hours of starting lenalidomide, and must either commit to continued abstinence from heterosexual intercourse or begin two acceptable methods of birth control, one highly effective method and one additional effective method at the same time, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counselled at a minimum of every 28 days about pregnancy precautions and risk of fetal exposure. Should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study, she should inform her treating physician immediately. FCBP must use adequate contraception for at least 28 days after discontinuation from study. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for at least 28 days after discontinuation from study
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients that have received prior IMiDs for treatment of ATLL
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who have not recovered to grade 1 or better from AEs due to prior anti-cancer therapy (not including cycle 1 of EPOCH, CHOP, or CHOPE if received off protocol) within 14 days prior to enrollment, with the exception of alopecia
* Patients who are receiving any other investigational agents or have received them within 14 days prior to enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lenalidomide or other agents used in study. Anaphylactic reactions including death have been reported with cyclophosphamide. Possible cross-sensitivity with other alkylating agents can occur
* Patients unable to take aspirin or prophylactic doses of low molecular weight heparin or direct oral anticoagulants
* Patients with urinary outflow obstruction (contraindication for cyclophosphamide)
* Patients with any form of demyelinating disease should not be given vincristine sulfate injection
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because lenalidomide is an IMiD agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lenalidomide, breastfeeding should be discontinued if the mother is treated with lenalidomide. These potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to the end of induction therapy
  Will determine the MTD for lenalidomide in combination with etoposide, prednisone, vincristine sulfate (Oncovin), cyclophosphamide, and doxorubicin hydrochloride (hydroxydaunorubicin hydrochloride) (EPOCH) chemotherapy.

SECONDARY OUTCOMES:
Overall response rate | Up to 2 years after completion of study treatment
  Will be summarized using descriptive statistics. Binomial proportions and their 95% confidence intervals will be used to estimate the response rates of therapy.
Duration of response | From the time measurement criteria are met for complete response (CR) or partial response (PR) until the first date that recurrent or progressive disease is objectively documented, assessed up to 2 years after completion of study treatment
  Will be summarized using descriptive statistics. The Kaplan-Meier method will be used to evaluate the response duration.
Progression-free survival | Up to 2 years after completion of study treatment
  Profession-free survival will be determined by the number of weeks from the time of initiation of therapy until there is evidence of tumor progression by acute T-cell leukemia (ATL) response criteria of Tuskasaki, 2009.
Overall survival | Up to 2 years after completion of study treatment
  Over survival will be determined by the number of week of weeks from the time of initiation of therapy until death.
T-cell receptor pathway gene mutational spectrum | Up to 2 years after completion of study treatment
  T-cell receptor pathway gene mutation will be determined by targeted next-generation sequence after hybridization to specific oligonucleotide capture probes corresponding to the sequence most commonly mutation in ATL as defined by Kataoka et al, 2015.
Human T-cell leukemia virus type 1 (HTLV-1) proviral deoxyribonucleic acid and ribonucleic acid loads | Up to 2 years after completion of study treatment
  Analysis of variance methods will be used to evaluate the effects of treatment and time on the viral load measurements, as well as measurements of viral transcripts.
HTLV-1 clonality | Up to 2 years after completion of study treatment
  HTLV-1 clonality will be determined by next generation sequence analysis of viral integration sites resulting in a distribution of the number of reads for each integration site plotted per integration site, as described by Gillet et al. 2011.
Incidence of toxicities | Up to the end of induction therapy
  The incidence of toxicities will be estimated using the binomial proportion and its 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ratner, Principal Investigator — Yale University Cancer Center LAO
Locations (19):
- United States (19):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm